CLINICAL TRIAL: NCT02685527
Title: Acute Gastroenteritis: Development of PCR Analysis and Algorithm/Criteria for Fast Clarification of Isolation Indication
Brief Title: Acute Gastroenteritis: Development of PCR Analysis and Algorithm for Fast Clarification of Isolation Indication
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: St. Franziskus Hospital (Other); Diakonissenkrankenhaus, Flensborg, Germany (Unknown); Aabenraa Hospital (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, associate professor, University of Southern Denmark
Other Study IDs: SHS-ED-02-2015
Record Dates: First submitted 2015-08-26; First posted 2016-02-18 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — feces for bacterial and virus determination
Oversight: Data Monitoring Committee: No

SUMMARY:
Isolation of contagious patients is expensive, requires more caregiver time, most of the patients perceive isolation as a mental strain and it has been shown that the level of care and observation is lower than in a normal ward. But isolation of contagious patients is necessary to protect other patients, hospital staff and relatives to prevent spreading of infection and, in worst case out-break.

There are different isolation regimes available depending on causative agent and mode of transmission. A community-acquired acute gastroenteritis (GE) is most often caused by Norovirus while a hospital-acquired acute GE is often caused by toxin producing Clostridium difficile. Patients infected with Norovirus or Clostridium difficile have to be isolated in single rooms with strict contact precautions. Patients infected with acute GE caused by other pathogens can be isolated in a multi-bed room if there is a private toilet.

However, at the time of arrival to hospital it is not known if the patient is contagious. The indication of isolation has to be made based of a clinical evaluation in risk of isolating to few or too many patients.

Aim of the study:

To identify anamnestic, clinical and paraclinical variables that can be used as indicators of the aetiology of infectious GE, thus giving an indication for isolation.

To clinically evaluate a combined RNA (Norovirus) and DNA (Clostridium difficile) fast PCR analysis test to identify infectious GE compared to gold standard methods.

ELIGIBILITY:
Inclusion Criteria:

* acutely admitted
* more than three Loose stool, or lest than three Loose stools and vomiting within the last three weeks

Exclusion Criteria:

* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted patients that contact an emergency department of the Hospital of Southern Denmark or St. Franziskus Hospital, Flensburg, Germany or Diakonissenkrankenhaus, Flensburg, Germany with symptoms of acute gastroenteritis.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
faeces examination for norovirus and clostridium difficile bacteria | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

REFERENCES:
- [Derived] Skyum F, Pedersen C, Andersen V, Chen M, Franke A, Petersen D, Ries W, Mogensen CB. Risk factors for contagious gastroenteritis in adult patients with diarrhoea in the emergency department - a prospective observational multicentre study. BMC Infect Dis. 2019 Feb 11;19(1):133. doi: 10.1186/s12879-019-3754-4. PMID 30744568